CLINICAL TRIAL: NCT05234918
Title: Comparative Evaluation of Two Different Paediatric Rotary File Systems and Manual K-file in Root Canal Treatment of Primary Teeth (Randomized Clinical Trial and In Vitro Study)
Brief Title: Evaluation of Different Paediatric Rotary Files and Manual K-file in Root Canal Treatment of Primary Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Huda Abd jabbar, Assisting teatcher, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED 21-1D
Record Dates: First submitted 2021-11-08; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Root Canal Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (Kedo S plus file study group) (Experimental): Group1: Kedo S plus file study group (The teeth will be instrumented by Kedo S plus file)
  Interventions: Device: Pediatric Rotary File Systems
- (Kidzo-file study group) (Experimental): Group2: Kidzo file study group (The teeth will be instrumented by Kidzo file)
  Interventions: Device: Pediatric Rotary File Systems
- (Manual K-file control group) (Experimental): Group3: Manual K-file control group (The teeth will be instrumented by Manual K-file)
  Interventions: Device: Pediatric Rotary File Systems

INTERVENTIONS:
Device: Pediatric Rotary File Systems — * Kedo S plus (p1 molar file ) (A1 anterior file)
  * Kidzo-file system 25/4 30/4 30/6

SUMMARY:
The aim of the current study is evaluation and comparsion between two different paediatric rotary file systems and Manual K-file both clinically and radiographically .This study consist of two parts:I-In vivo part (RCT) II-In vitro part

The in-vivo part:

Its sample size was found to be 30 primary molars (10 teeth for each group)

Group1: Kedo S plus file study group (The teeth will be instrumented by Kedo S plus file) Group2: Kidzo file study group (The teeth will be instrumented by Kidzo file) Group3: Manual K-file control group (The teeth will be instrumented by Manual K-file)

Pulpectomy of primary molars according the protocol of individual group will be made, after that the teeth will be evaluated Immediately for :

1-Instrumentation time 2-Quality of obturation and evaluated at 1, 3, 6, 12 months for clinical and radiographic success

DETAILED DESCRIPTION:
The aim of the current study is to evaluation and comparsion between two different paediatric rotary file systems (Kedo S plus file and Kidzo File) and Manual K-file both clinically and radiographically

Primary Objective:

Evaluation of clinical success, instrumentation time and quality of obturation of two different paediatric rotary file systems and manual K-file system in pulpectomy in primary molars both clinically and radiographically (In-vivo part of the study).

Testing hypothesis:

The null hypothesis (H 0 ): there is no difference in clinical success, instrumentation time ,quality of obturation and apical debris extrusion between the two different pediatric rotary systems and manual K-file system in pulpectomy in primary molars

PICOTS:

P - Participants: Children in the age group of 4-7 years having pulpally involved Primary teeth indicated for pulpectomy, I - Intervention: Pulpectomy procedure in primary molars using Kedo S plus file and Kidzo file.

C - Comparison: Manual K-file.

O- Outcomes:

* Clinical and Radiographic success
* Instrumentation time T- Clinical and radiographic follow up over 12-month period. S- Randomized clinical trial (RCT) and in-vitro study.

The predicted sample size was found to be 30 teeth (10 teeth per group) which was calculated by using G*Power version 3.1.9.7. Sample size will be increased by about 10% to compensate for the drop out.

Selection of primary molars, of 4 to 7 year old patients, following the inclusion criteria N=30

All Participant will be a randomly allocated into one of the either group (10 teeth in each group):

Group1: Kedo S plus file study group (The teeth will be instrumented by Kedo S plus file) Group2: Kidzo file study group (The teeth will be instrumented by Kidzo file) Group3: Manual K-file control group (The teeth will be instrumented by Manual K-file)

Pre-operative intraoral periapical radiograph for assessing the root structure and confirming the diagnosis of pulpal involvment

Pulpectomy of primary molars according the protocol of individual group

• Materials and Clinical procedures

In this study, the following materials will be used:

* Manual K-file
* Two different rotary paediatric file
* Endomotor with apexolocator
* Calcium hydroxide with iodoform paste
* Polymer Reinforced ZOE Cement (IRM)
* Glass Ionomer Cement
* Stainless Steel Crown Clinical procedure Group 1: (Kedo S plus file study group)

  1. Pre-operative Intra Oral Periapical radiograph of the teeth will be taken using the standardized paralleling technique .
  2. Topical and local anesthesia will be administered.
  3. Tooth will be isolated with rubber dam.
  4. Caries will be removed.
  5. The convenience access will be with reached by a carbide bur without active tip (Endo Z).
  6. The canal orifices will be localized with a #10 hand K-file.
  7. The working length will be determined using the apex locator with one mm shorter than the '0.0' mark in apex locator.
  8. Kedo S plus file will be used for instrumentation according to manufacturer's instructions.
  9. Between the use of each file, the canals will be irrigated with sodium hypochlorite and EDTA gel "17%" will be used for lubrication of files during instrumentation.
  10. Canals will then be dried with sterile paper points .
  11. Metapex will then be administrated into the canals using pressure syringe technique followed by final compaction of the material by using wet cotton pellets technique.
  12. The access cavity will be restored by Zincinol
  13. Final coronal restoration of the pulpectomized tooth will be achieved using a preformed stainless steel metallic crown luted with glass ionomer cement.
  14. Immediate postoperative intraoral periapical radiograph will beobtained for assessment of quality of obturation.

Group 2: (Kidzo-file study group) Steps 1-7 will be done as mentioned above. Then, Kidzo file will be used for instrumentation according to manufacturer's instructions. Step 9-14 also, will be repeated as well.

Group 3: (Manual K-file control group) Steps 1-7 will be done as mentioned above also. Then, the teeth will be instrumented by using hand k-files. Again step 9-14 will be repeated as well.

* Follow-up The patients will be recalled for clinical and radiographic follow up after 1, 3, 6 and 12 months.
* Outcome measurement

  1. Immediate post operative

     A-The instrumentation time:

     Will be recorded using a digital stopwatch, which include only instrumentation time of the used files excluding the in-between irrigation protocol for assessing the accurate time period needed for instrumentation in each group.

     B-The quality of obturation:

     Will be assessed according to criteria of Coll and Sadrian (1996) as (Underfilled, Optimal filled or Overfilled) by using intraoral periapical radiograph by paralleling technique.
  2. Through the follow up period:

  <!-- -->

  1. Clinical and radiographic success The following table indicating to the clinical and radiographic Coll and Sadrian.

     criteria for treatment success,(1996) (44) : Clinical criteria Radiographic criteria 1. Absence of pain on percussion on recall checkup 1. No pathologic root resorption 2. No gingival swelling or sinus tract 2. No widening of the periodontal ligament space 3. Absence of purulent exudate expressed from the gingival margin 3. Absence or decrease of any periapical or furcation involvement 4. No abnormal mobility of tooth
* Blinding Participants and legal guardian will be blinded to which group they will be allocated , and the evaluator also will be blinded. While the operator /primary investigator cannot be blinded as she is already familiar with the type of the files used and their different instruction for using. For statistical analysis, codes will also assure blinding and confidentiality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the age of 4-7 years.
2. Posterior primary mandibular molars with necrotic pulp or irreversible pulpitis indicated for pulpectomy .
3. Presence of minimum 2/3rd root structure.
4. Adequate restorable tooth structure for further placement of stainless steel crowns.
5. Medically free patient.
6. Patient able to visualize and understand the explained assent with no impairment.

Exclusion Criteria:

1. Teeth of poor prognosis due to presence of an extensive mobility, advanced bone or root resorption.
2. Uncooperative patient
3. parents who refuse to sign informed consent to participate in the study

   -

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
clinical outcome through participant clinical examination | from baseline to 12 months
  Evaluation of participants with clinical success according to Coll and Sadrian criteria for treatment success No pain, No sweeling , No exudate, No abnormal mobility
The quality of obturation will be assessed by using periapical intra oral radiographic parallel technique | from baseline to 12 months
  the quality of obturation will be assessed from the obtained x - ray film by visual examination to evaluate it under the following categories: Under filled- Optimal filled- Over filled
Instrumentation time | immediatly after procedure
  time of instrumentation will be measured immediatly by digital watch in seconds

IPD SHARING:
Plan to Share IPD: No